CLINICAL TRIAL: NCT04812418
Title: Evaluation of a Combination of Plants in Anxiety-related Sleep Disorders: Randomized Trial Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Organization: Larena SAS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pil-Clin-Noct-020
Record Dates: First submitted 2021-01-15; First posted 2021-03-23 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Sleep Troubles Associated With Anxiety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): 120 mg of eschscholtzia extract and 50 mg of valerian extract by tablet, without support 28 days
  Interventions: Dietary Supplement: Noctesia
- Group (B) (Placebo Comparator): Placebo 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Noctesia — 3 tablets every day at bedtime with a large glass of water
  Arms: Group (A)
Dietary Supplement: Placebo — 3 tablets every day at bedtime with a large glass of water
  Arms: Group (B)

SUMMARY:
The objective of this double-blind randomized clinical trial is to compare the effects of a dietary supplement based on eschscholtzia and valerian extracts to a placebo after 28 days of supplementation, in subjects suffering from sleep troubles associated with anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man, aged of 18 to 65 years;
* In good general health as evidenced by medical history and physical examination;
* Having at least 3 episodes of sleep disorders per week including one or more of the following:

  1. difficulty falling asleep or
  2. difficulty staying asleep or
  3. poor quality sleep
  4. Waking up earlier than desired
* The insufficient sleep duration and quality is coupled with a feeling of general fatigue;
* Sleep disorder last for more than 1 month;
* Presenting moderate to severe sleep disorder in the past month (ISI ≥ 15);
* With anxiety resulting in a HAM-A score > 8 and < 25;
* For women of childbearing age (women of childbearing potential, pre-menopausal or having postmenopausal amenorrhea of less than 12 months, and women who have not undergone surgical sterilization):

  1. Negative blood pregnancy test
  2. Acceptance to use an effective method of contraception, established for at least 1 month, and throughout the duration of the study;
* Fluent French speaking;
* Provision of signed and dated informed consent form;
* Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* A score > 10 on the ESS scale (that would correspond to serious hypersomnia);
* Sleep disorders secondary to another health problem (sleep apnea syndrome, narcolepsy-cataplexy, idiopathic hypersomnia, restless legs syndrome, chronic pain syndrome, ...) or an environmental factor (noise, light ...) or socio-professional (shift work, young child at home, people who are often jet lagged,… );
* Severe psychiatric disorder or disease within 6 months before inclusion (depression, bipolar disorder, severe anxiety, psychosis, schizophrenic disorders, dementia,…) or a severe neurologic trouble (Alzheimer's, autism, Parkinson's disease, …);
* Subjects presenting severe gastro-intestinal, hepatic, respiratory, kidney or cardiovascular disorder or severe infection (e.g. HIV, hepatitis, …);
* Acute or chronic somatic pathologies which can interfere with sleep: kidney cancer, etc.;
* Subjects with pre-menstrual syndrome or myasthenia gravis;
* Subjects who drink more than 2 glasses of alcohol per day (> 20g of alcohol per day) or with exaggerated consumption of theine (≥ 1l per day) and caffeine-rich (≥ 800ml per day) beverages and energy drink (≥ 330ml per day);
* Smoker;
* Subject consuming drugs and/or with historical drug addiction;
* Under psychotropic treatment within the last month before screening (neuroleptic, anxiolytic, antidepressant, hypnotic, sedative, …) or under current medication treatment which may alter the waking state (for example: cortisone, dopamine, amphetamine, antihistamines, beta-blockers, certain cough syrups, .…);
* Volunteer with suicidal risk according to the investigator;
* Under phytotherapy treatment or food supplement for sleep disorders within the last month before screening;
* Volunteer presenting current infection and/or fever;
* Volunteer with medical history of stroke or head trauma;
* Pregnant or lactating woman;
* Known allergy or intolerance to one product component (valerian, eschscholtzia or excipients);
* Subjects having participated to another clinical trial (with an investigational product) one month before the inclusion;
* Subjects that present alterations of their cognitive functions that will interfere with the comprehension of the study and procedures and/or with the completion of questionnaires;
* Vulnerable patient (deprived of liberty by judicial or administrative decision, under guardianship, curatorship or safeguard of justice, …);
* Pharmacological resistance to common hypnotic/sedative drugs;
* Allergy/intolerance to the actimeter straps;
* Recent (< 1 month before the inclusion) change in lifestyle (food, body weight > 5kg, sport).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Sleep disorder severity | Baseline and D28 (end of supplementation)
  Change from baseline of Insomnia Severity Index (ISI) score

SECONDARY OUTCOMES:
Sleep disorder severity over time | Baseline and D49 (end of follow-up)
  Change from baseline of Insomnia Severity Index (ISI) score
Investigator assessment of sleep disorder symptoms severity | Baseline and D28 (end of supplementation)
  Change from baseline of Clinical Global Impression Severity (CGI-S) score
Investigator assessment of sleep disorder symptoms improvement | Baseline and D28 (end of supplementation)
  Change from baseline of Clinical Global Impression Improvement (CGI-I) score
Patient assessment of sleep disorder symptoms improvement after intervention | Baseline and D28 (end of supplementation)
  Change from baseline of Patient Global Impression Improvement (PGI-I) score
Anxiety status | Baseline and D28 (end of supplementation)
  Change from baseline of Hamilton anxiety rating scale (HAM-A) score
Anxiety status over time | Baseline and D49 (end of follow-up)
  Change from baseline of Hamilton anxiety rating scale (HAM-A) score
Short-form 36 questionnaire (SF36) | Baseline and D28 (end of supplementation)
  Change from baseline of SF36 scores
Actimeters | Baseline, D7, D14, D21 and D28 (end of supplementation)
  Change from baseline of the mean values obtained from actimeters recording during the 7 days
Electronic sleep diaries | Baseline, D7, D14, D21 and D28 (end of supplementation)
  Change from baseline of the mean values obtained from electronic sleep diaries during the 7 days
Evolution of sleep troubles | Baseline, D28 (end of supplementation) and D49 (end of follow-up)
  Change from baseline of sleep troubles regarding changes in medical prescriptions, reason of changes and number of intercurrent medical visits for sleep disorders
Addiction | Baseline and D49 (end of follow-up)
  Change from baseline of Addiction questionnaire scores
Adverse events | Baseline D7, D14, D21, D28 (end of supplementation) and D49 (end of follow-up)
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique en Nutrition, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No